CLINICAL TRIAL: NCT03287362
Title: The OPTIMA-Study: Optimized Treatment Identification at the Max Planck Institute of Psychiatry
Brief Title: Effects of Schema Therapy vs. Cognitive Behavioral Therapy vs. Individual Supportive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-395
Record Dates: First submitted 2017-08-25; First posted 2017-09-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; cognitive behavioral therapy; supportive therapy; schema therapy; biomarkers; neuropsychology; circadian rhythm
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Schema Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Incoming patients from the clinic of Max Planck Institute of Psychiatry are continuously screened for study eligibility and - after they have given informed consent - are block wise randomly assigned to one of 3 study arms (schema therapy, cognitive behavioral therapy, individual supportive therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ST-arm (Experimental): one-third of the patients is randomized to schema therapy
  Interventions: Behavioral: schema therapy
- CBT-arm (Active Comparator): one-third of the patients is randomized to cognitive behavioral therapy
  Interventions: Behavioral: cognitive behavioral therapy
- IST-arm (Placebo Comparator): one-third of the patients is randomized to individualized supportive therapy
  Interventions: Behavioral: individualized supportive therapy

INTERVENTIONS:
Behavioral: schema therapy — The intervention consists of a seven-week program of schema therapy, which is a further development of cognitive behavioral therapy, designed in a three-phase combined group and single session concept
  Arms: ST-arm
Behavioral: cognitive behavioral therapy — The intervention consists of a seven-week program of cognitive behavioral therapy, which is the current gold standard of treatment
  Arms: CBT-arm
Behavioral: individualized supportive therapy — The intervention consists of a seven-week program of individualized supportive therapy, including different therapeutic offers from the clinic and a high frequency of physician contacts.
  Arms: IST-arm

SUMMARY:
The OPTIMA-Study: Optimized Treatment Identification at the Max Planck Institute of Psychiatry: An outline

Depressive disorders represent one of the most frequent diseases worldwide. Schema therapy, which was originally developed for patients with personality disorders and focuses on emotion activating techniques, became popular in the field of psychotherapy in the recent years and was also applied on axis-I-disorders such as depression.

The current study aims to close the gap of increasing popularity of ST and missing empirical evidence of its effectiveness. This aim breaks down into three main research questions dealing with (1) general effectiveness of ST measured by multiple operationalizations (i.e. depressive symptoms, biological markers, relapse prevention, or need for medication), (2) specific effectiveness of ST (i.e. interpersonal problems and emotion regulation), and (3) the identification of parameters in the sense of an individualized psychotherapy approach in order to fit patient needs with certain psychotherapy offers.

After participants have given informed consent, they undergo a comprehensive baseline measurement which covers psychometric measures (such as questionnaires and clinical ratings), biological parameters (blood samples, endocrine activity), neuropsychological testing (such as word fluency), and actimetry measures (circadian rhythms).

After finishing the diagnostic procedure, participants will be randomized to three different experimental conditions: (1) a schema therapy condition, (2) a cognitive behavioral therapy condition, and (3) an individualized supportive therapy condition. After undergoing a comprehensive baseline measurement process in study week one, patients participate in an intensive seven-week-treatment-program, in addition to the regular pharmacological treatment, which is not object of the study. The measures are repeated during the fourth and seventh week of psychotherapeutical treatment and on the occasion of a follow-up visit six months after discharge from the clinic.

Additionally, the investigators test among sub-samples the effects of psychotherapeutical interventions on psychophysiological outcomes, sleep-patterns, and neuronal substrates in the context of emotional regulation and social interaction.

Thus, the study will give valuables insights in the effectiveness of an innovative psychotherapy approach and breaks new ground in the field of individualized psychotherapy and its biological implications.

ELIGIBILITY:
Inclusion Criteria:

1. Main diagnosis of major depressive disorder, single episode or recurrent, moderate or severe without psychotic symptoms according to DSM-5 criteria (F32.1, F32.2, F33.1, F33.2 according to ICD-10)
2. age between 18 and 75 years
3. informed consent to the study procedures and assessments (in written form)

Exclusion Criteria:

1. Major depressive disorder, single episode or recurrent, severe with psychotic symptoms (F32.3, F33.3 according to ICD-10)
2. Severe mutism or stupor
3. lifetime history of any psychotic or bipolar disorder
4. severe neurological or internal concomitant diseases
5. IQ < 80; severe learning disability, brain damage or pervasive developmental disorder
6. current alcohol or any illicit drug withdrawal syndrome according to DSM-5
7. mental disorders secondary to a medical conditions or substance use disorders
8. acute suicidality
9. pregnancy and lactation period
10. Missing eligibility for psychotherapy because of missing language skills
11. Electroconvulsive therapy (ECT) in preparation
12. Participation in further scientific studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
BDI-II (Beck-Depression-Inventory-II) | Assessed as baseline measure after informed consent was given, and on a weekly base over the course of seven weeks of treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Decrease in depression symptoms, measured by "benefit" changes in scores of BDI-II (Beck-Depression-Inventory-II) questionnaire (self rating) from baseline over the course of seven weeks of treatment up to six months after discharge from the clinic

SECONDARY OUTCOMES:
MADRS (Montgomery-Åsberg Depression Rating Scale) | Assessed as baseline measure after informed consent was given, in week 4 and 7 of the treatment.Additionally in a follow-up assessment six months after discharge from the clinic.
  Decrease in depression symptoms, "benefit" changes from baseline to week 4 and 7 of treatment up to six months after discharge from the clinic, clinical rating
CIDI (Composite International Diagnostic Interview) | Assessed as baseline measure after informed consent was given, in week 7 of the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Decrease in symptoms or recovery from DSM-5 diagnosis of depression, "benefit" changes from baseline to week 7 of treatment and up to six months after discharge from the clinic
BSI (Brief Symptom Inventory) | Assessed as baseline measure after informed consent was given, and on a weekly base over the course of seven weeks of treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Decrease in general psychopathology, "benefit" changes from baseline over the course of seven weeks of treatment up to six months after discharge from the clinic
WHOQOL (WHO - Quality of Life) | Assessed as baseline measure after informed consent was given, in week 4 and 7 of the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Increase in quality of life, "benefit" changes from baseline to week 4 and 7 of treatment and up to six months after discharge from the clinic
Neuropsychological testing (including sections on episodic memory, working memory, inhibition, cognitive flexibility, word fluency, sensitivity to interference, and attention) | Assessed as baseline measure after informed consent was given, in week 4 and 7 of the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Increase of cognitive functioning, "benefit" changes from baseline to week 4 and 7 of treatment and up to six months after discharge from the clinic
Decreased need for psychopharmacological medication | Comparison between baseline measurement before treatment start and end of therapy treatment of seven weeks
Dropout rate from therapeutic treatment | Assessed after all participants were recruited, enrolled, treated and finished their final measurements (approx. after eight years)
WHODAS (WHO-Disability Assessment Schedule) | Assessed as baseline measure after informed consent was given, in week 7 of the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Decrease in symptoms or recovery from DSM-5 diagnosis of depression, "benefit" changes from baseline to week 7 of treatment and up to six months after discharge from the clinic

OTHER OUTCOMES:
PID-5 | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  The Personality Inventory for DSM-5
YSQ-S2 | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment.. Additionally in a follow-up assessment six months after discharge from the clinic.
  Young Schema Questionnaire
ATQ | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Automatic Thought questionnaire
DAS | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Dysfunctional Attitude Scale
NAQ | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Need for Affect Questionnaire
IE-4 | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  a short scale to assess internal and external control beliefs
ERQ | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Emotion Regulation Questionnaire
RSQ-D | Assessed as baseline measure after informed consent was given and in week 7 after finishing the treatment. Additionally in a follow-up assessment six months after discharge from the clinic.
  Response Styles Questionnaire
MCTQ | Assessed in week 4.
  Munich ChronoType Questionnaire
blood samples | Assessed as baseline measure after informed consent was given, in week 4 and 7 of the treatment.Additionally in a follow-up assessment six months after discharge from the clinic.
endocrine parameters | Assessed as baseline measure after informed consent was given, in week 4 and 7 of the treatment.
ECG | Assessed at baseline and in week 7.
circadian rhythms | continuous measurement using a wearable actimeter during the whole therapy program of seven weeks
imaging (MRT) | Assessed at baseline and in week 7.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes M. Kopf-Beck, PhD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renner F, van Goor M, Huibers M, Arntz A, Butz B, Bernstein D. Short-term group schema cognitive-behavioral therapy for young adults with personality disorders and personality disorder features: associations with changes in symptomatic distress, schemas, schema modes and coping styles. Behav Res Ther. 2013 Aug;51(8):487-92. doi: 10.1016/j.brat.2013.05.011. Epub 2013 May 31. PMID 23778056
- [Background] Ferrari AJ, Charlson FJ, Norman RE, Patten SB, Freedman G, Murray CJ, Vos T, Whiteford HA. Burden of depressive disorders by country, sex, age, and year: findings from the global burden of disease study 2010. PLoS Med. 2013 Nov;10(11):e1001547. doi: 10.1371/journal.pmed.1001547. Epub 2013 Nov 5. PMID 24223526
- [Derived] Kirchler SV, Muller CL, Spock Z, Ehring T, Kopf-Beck J, Tamm J. The role of concreteness in repetitive negative thinking: Temporal dynamics and the predictive value for depression throughout psychological treatment. Behav Res Ther. 2025 Sep;192:104801. doi: 10.1016/j.brat.2025.104801. Epub 2025 Jun 11. PMID 40544720
- [Derived] Tamm J, Takano K, Just L, Ehring T, Rosenkranz T, Kopf-Beck J. Ecological Momentary Assessment versus Weekly Questionnaire Assessment of Change in Depression. Depress Anxiety. 2024 Jul 11;2024:9191823. doi: 10.1155/2024/9191823. eCollection 2024. PMID 40226649
- [Derived] Kopf-Beck J, Muller CL, Tamm J, Fietz J, Rek N, Just L, Spock ZI, Weweck K, Takano K, Rein M, Keck ME, Egli S. Effectiveness of Schema Therapy versus Cognitive Behavioral Therapy versus Supportive Therapy for Depression in Inpatient and Day Clinic Settings: A Randomized Clinical Trial. Psychother Psychosom. 2024;93(1):24-35. doi: 10.1159/000535492. Epub 2024 Jan 4. PMID 38176391
- [Derived] Kopf-Beck J, Zimmermann P, Egli S, Rein M, Kappelmann N, Fietz J, Tamm J, Rek K, Lucae S, Brem AK, Samann P, Schilbach L, Keck ME. Schema therapy versus cognitive behavioral therapy versus individual supportive therapy for depression in an inpatient and day clinic setting: study protocol of the OPTIMA-RCT. BMC Psychiatry. 2020 Oct 14;20(1):506. doi: 10.1186/s12888-020-02880-x. PMID 33054737